CLINICAL TRIAL: NCT04429373
Title: Effect of Platelet-rich Plasm (PRF) on Two-implant Mandibular Overdenture: a Split Mouth
Acronym: PRF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Franco Cavalla, Assistant Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ORF42004
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Edentulous Jaw; Dental Implant Failed
Keywords: dental implants; platelet-rich plasm; edentulous jaw
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Intervention Model Description: We will conduct a split-mouth design randomized clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Allocation sequence will be masked from participant, outcome assessor and statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implant installation with PRF (Experimental): PRF membrane over the buccal aspect of implant site
  Interventions: Procedure: Implant installation with PRF membrane
- Implant installation without PRF (Active Comparator): Implant installation contralateral to the the experimental implant, without PRF membrane
  Interventions: Procedure: Implant installation without PRF membrane

INTERVENTIONS:
Procedure: Implant installation with PRF membrane — Platelet-rich fibrin membrane over the buccal aspect of implant site after dental implant installation
  Arms: Implant installation with PRF
Procedure: Implant installation without PRF membrane — Implant installation contralateral to the experimental side without PRF membrane
  Arms: Implant installation without PRF

SUMMARY:
Implant retained overdentures are a cost-effective treatment for elderly patients suffering from complete tooth loss. Despite the high success rate of implants in the general population, older adults lacking all teeth are a challenging population for implant therapy, often presenting limited bone disponibility, narrow alveolar ridges, diminished bone density, scarce inserted gingiva and several co-morbidities.Thus, improving their possibility of success in implant therapy avoiding further surgical interventions is key.

Platelet-rich fibrin (PRF) is a blood derivate that can be easily and economically obtained from patients and that has shown promise of reducing the complications and improving the success of implant therapy, nevertheless its benefits in patients receiving implant retained overdentures has not been stablished. It is possible that PRF can improve the results and diminish the complications of implant therapy in older adults.

The investigation aims to demonstrate that the use of platelet-rich fibirn (PRF) is safe and beneficial for implant treatment in older adults suffering from complete tooth loss.

DETAILED DESCRIPTION:
The investigators will conduct a split-mouth design randomized clinical trial assessing the effect of PRF in primary stability and bone/soft tissue healing around mandibular implants in edentulous elderly adults.

Aim and purpose

1. To assess the effect of PRF on primary implant stability of mandibular implants in edentulous patients using resonance frequency analysis (RFA).
2. To evaluate the effect of PRF on clinical parameters related to soft tissue healing, post-surgical pain/inflammation and early complications of mandibular implants in edentulous patients.
3. To examine soft tissues volumetric changes pre and post- surgery using intraoral scans and bone changes using cone-beam computed tomography (CBCT) around mandibular implants in edentulous patients.

ELIGIBILITY:
Inclusion Criteria:

* mandibular edentulous
* > 60 years old

Exclusion Criteria:

* physical or psychological impediment for dental surgery
* dental extraction < 6 months in the mandible
* anticoagulant treatment

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Implant stability | 6 months
  primary implant stability of mandibular implants in edentulous patients using resonance frequency analysis (RFA).

SECONDARY OUTCOMES:
Keratinized tissue thickness around implant neck | 6 months
  Distance in mm from the surface of keratinized gingiva 1 mm apical to implant neck to bone contact
Keratinized tissue width around implant neck | 6 months
  Distance in mm of keratinized tissue from implant neck to mucogingival junction

CONTACTS AND LOCATIONS:
Locations (1):
- San Camilo Hospital, San Felipe, Aconcagua, Chile

IPD SHARING:
Plan to Share IPD: No